CLINICAL TRIAL: NCT02458014
Title: Phase II Study of Blinatumomab in Patients With B-Cell Lineage Acute Lymphocytic Leukemia With Positive Minimal Residual Disease
Brief Title: Blinatumomab in Treating Patients With B-cell Acute Lymphoblastic Leukemia With Minimal Residual Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0844; NCI-2015-01547 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0844 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-05-26; First posted 2015-05-29 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Adult Acute Lymphoblastic Leukemia in Complete Remission; B Acute Lymphoblastic Leukemia; Minimal Residual Disease; Philadelphia Chromosome Positive
MeSH Terms: conditions — Burkitt Lymphoma; Neoplasm, Residual | interventions — blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (blinatumomab) (Experimental): Patients receive blinatumomab IV continuously on days 1-28. Treatment repeats every 6 weeks for up to 5 courses in the absence of disease progression or unacceptable toxicity. Patients who do not proceed with stem cell transplantation may receive blinatumomab IV maintenance therapy with one cycle every 3 months for up to 4 cycles. Patients who remain in MRD remission for 3 months and then become MRD positive again can be retreated following the same treatment plan previously received.
  Interventions: Biological: Blinatumomab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Blinatumomab — Given IV
  Other Names: Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI-538; MT-103
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well blinatumomab works in treating patients with B-cell acute lymphoblastic leukemia whose disease is in remission (causes no symptoms or signs) but is still present in a small number of cells in the body (minimal residual disease). Immunotherapy with monoclonal antibodies, such as blinatumomab, may induce changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the clinical efficacy of blinatumomab in patients B-cell acute lymphoblastic leukemia in complete morphologic remission with positive minimal residual disease (MRD) in terms of relapse-free survival (RFS).

SECONDARY OBJECTIVES:

I. To evaluate other efficacy endpoints such as overall survival and MRD negativity rate by flow cytometry and/or polymerase chain reaction (PCR) overall and after the first cycle, as well as safety of blinatumomab in this setting.

OUTLINE:

Patients receive blinatumomab intravenously (IV) continuously on days 1-28. Treatment repeats every 6 weeks for up to 5 cycles in the absence of disease progression or unacceptable toxicity. Patients who do not proceed with stem cell transplantation may receive blinatumomab IV maintenance therapy with one cycle every 3 months for up to 4 cycles. Patients who remain in MRD remission for 3 months and then become MRD positive again can be retreated following the same treatment plan previously received.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with B-lineage acute lymphocytic leukemia (ALL) in hematologic complete remission (CR) with molecular failure (i.e., had never achieved an MRD-negativity status before blinatumomab) or had a molecular relapse (i.e., became MRD positive after having been MRD negative) starting at any time point after 3 months of frontline therapy; molecular disease or minimal residual disease is defined by a value of at least of 1 x 10^-4 (0.01%) by multicolor flow cytometry and/or by next generation sequencing (NGS)
* Patients with B-lineage ALL in hematologic complete remission (CR) with molecular failure (i.e., had never achieved an MRD-negativity status before blinatumomab) or had a molecular relapse (i.e., became MRD positive after having been MRD negative) starting at any time point after 3 months of frontline therapy; molecular disease or minimal residual disease is defined by a value of at least of 1 x 10-4 (0.01%) by multicolor flow cytometry and/or by next generation sequencing (NGS)
* Performance status of 0, 1, or 2
* Creatinine clearance >= 30 ml/minute
* Bilirubin less than or equal to 3.0 mg/dL
* No active or co-existing malignancy with life expectancy less than 12 months
* Patients with Philadelphia chromosome positive (Ph+) ALL can be enrolled in CR1 or CR2 and beyond; a tyrosine kinase inhibitor (TKI) will be added at the discretion of the treating physician; MRD for these patients will be defined by PCR of 0.1% and above (International Scale)

Exclusion Criteria:

* Pregnant or nursing women
* Known to be human immunodeficiency virus positive (HIV+)
* Active and uncontrolled disease/infection as judged by the treating physician
* Unable or unwilling to sign the consent form
* Active central nervous system (CNS) or extramedullary disease
* Monoclonal antibodies therapy within 2 weeks before study entry
* Radiotherapy and cancer chemotherapy (except for intrathecal prophylaxis and/or low-dose maintenance therapy such as vinca alkaloids, mercaptopurine, methotrexate, steroids) or any investigational drug within 2 weeks before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | From date of treatment start until the date of death or hematologic or extramedullary disease relapse, assessed up to 18 months
  RFS will be estimated using the method of Kaplan and Meier. Will compute the Bayesian posterior probability. As a secondary analysis, will perform a competing risk analysis treating stem cell transplant as a competing event for RFS. In addition, will assess the RFS in the subgroup of patients with minimal residual disease (MRD) positivity in at least marrow complete remission (CR) 2 beyond, or in the subgroup of patients with and without allogenic stem cell transplant (ASCT), if permitted by the sample size. Landmark analysis may be performed to assess the difference in RFS between patients with or without receiving ASCT, if permitted by the sample size.

SECONDARY OUTCOMES:
Event-free survival | Up to 18 months
  Defined as RFS in addition to lack of achievement of negative MRD status after 2 cycles of blinatumomab (events will include death, lack of response after 2 cycles, and loss of response/progression, including MRD recurrence).
Overall survival (OS) | Up to 18 months
  OS will be estimated using the method of Kaplan and Meier. Will assess OS in the subgroup of patients with MRD positivity in at least marrow CR 2 beyond; or in the subgroup of patients with and without ASCT, if permitted by the sample size. Landmark analysis may be performed to assess the difference in OS between patients with or without receiving ASCT, if permitted by the sample size.
MRD negativity rate | Up to 18 months
  Will be estimated along with the exact 95% confidence interval.
MRD negativity rate after course 1 | Up to 6 weeks
  Will be estimated along with the exact 95% confidence interval.
Incidence of toxicity | Up to 18 months
  All treated patients are included in the safety analysis set. The adverse events will be summarized by organ type, grade and attribution to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jabbour EJ, Short NJ, Jain N, Jammal N, Jorgensen J, Wang S, Wang X, Ohanian M, Alvarado Y, Kadia T, Sasaki K, Garris R, Garcia-Manero G, Ravandi F, Kantarjian HM. Blinatumomab is associated with favorable outcomes in patients with B-cell lineage acute lymphoblastic leukemia and positive measurable residual disease at a threshold of 10-4 and higher. Am J Hematol. 2022 Sep;97(9):1135-1141. doi: 10.1002/ajh.26634. Epub 2022 Jun 24. PMID 35713551
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT02458014/ICF_000.pdf